CLINICAL TRIAL: NCT01527435
Title: Zeaxanthin as an Adjuvant to Combination Therapy for Treatment of Choroidal Neovascularization (CNV) in Exudative Age Related Macular Degeneration (ARMD)
Brief Title: Addition of 20mg/Day Zeaxanthin to Triple Therapy Treatment Options for Age Related Macular Degeneration (ARMD)
Acronym: ARMD
Status: Completed | Type: Observational
Sponsor: The Retina Center of St. Louis County, PC (Other)
Collaborators: ZeaVision, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 11-06-0044
Record Dates: First submitted 2012-01-27; First posted 2012-02-07 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Exudative Age-Related Macular Degeneration
Keywords: Best corrected visual acuity; Slit lamp examination; Ophthalmoscopy with contact lens/indirect ophthalmoscope; OCT assessment; Fundus photos, fluorescein angiogram, ICG angiogram

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the fact that 20 milligrams per day of oral Zeaxanthin as a supplement to patients with Choroidal neovascularization (CNV) and exudative age related macular degeneration (ARMD) undergoing combination therapy with intravitreal Bevacizumab (Avastin), intravitreal Dexamethasone and PDT laser photocoagulation and improves anatomic and visual outcome compared to patients not receiving oral Zeaxanthin. Study patients will be taking AREDS(PreserVision) and multivitamins (Centrum Silver); in addition one-half of the patients will receive 20mg of oral Zeaxanthin.

DETAILED DESCRIPTION:
One of the current treatments for choroidal neovascularization in exudative age related macular degeneration (ARMD) involves a combination of laser photocoagulation (PDT) and injections of an anti-inflammatory (Dexamethasone) and an anti-angiogenic (Bevacizumab). This combination therapy is designed to stabilize vision, improve vision in selected cases and reduce the total number of treatment cycles overall compared to other methods of treatment presently in use. Many retinal physicians are treating exudative ARMD with an ocular injection every 4 weeks for a number of years. Combination therapy has reduced the number of treatment cycles to less than 3 for many patients; and in preliminary studies, patients taking 20 milligrams of dietary oral zeaxanthin required even less treatment cycles to achieve stability. In this trial, the only variable will be the oral consumption of 20 milligrams of zeaxanthin daily taken in half of the patients randomized to this group. The remaining half patients with still undergo combination therapy, but without taking 20 milligrams of oral dietary Zeaxanthin.

Zeazanthin is found in many foods and low doses of zeazanthin are commonly added to many multivitamins already on the market. All products with Zeazanthin is a constituent, including EyePromise Ten, have excellent safety profiles and no side effects or adverse events have been reported thus far with this supplement.

Zeazanthin is in many eye supplements and is being studied by the NEI, National Eye Institute, as part of the AREDS-2 study looking at the benefits of Lutein, Zeazanthin and Omega 3 Fish Oils on AMD progression. The patients will be taking 20 milligrams a day of Zeazanthin. The United States and global safety organization have established an ADI (acceptable daily intake) of 2 mg/kg body weight/day of Zeazanthin. This equates to 155 mg per day for 177 pound person.

Millions of doses of EyePromise Ten have been taken without side effects. The new part of this trial, again is taking 20 milligrams of Zeazanthin while being combined with medical injections and laser treatments. Zeazanthin is one of the two pigments obtained from the diet that deposit in the macula and give it the yellow color. While obtained from the diet the retina accumulates it up to 1000 times higher levels than anywhere else in the body. Numerous scientific and clinical trials suggest that it is critical to the protection of the retina and in reducing risks and progression of age related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female at least 50 years of age.
2. Subjects must have age related macular degeneration with a choroidal neovascular membrane either classic or occult in at least one eye.
3. Preoperative best corrected visual acuity (BCVA) equal to or greater to 19 letters on the ETDRS diabetic retinopathy study chart (20/400 Snellen).
4. Media clarity, pupillary dilation and subject cooperation sufficient for accurate OCT and angiographic assessment.
5. Written and informed consent has been obtained.
6. Written authorization for the use and release of the health and research study information in the United States of America USA.
7. Ability to understand the informed consent and willingness to follow study instruction and likely to complete all required visits and procedures.

Exclusion Criteria:

1. Evidence of diabetic retinopathy or other retinal disease other than age related macular degeneration.
2. Any severe active ocular disease or condition that in the opinion of the investigator is severe enough to prevent a 3 line improvement in visual acuity or to compromise the study results.
3. Any presumed ocular infections, i.e. bacterial, viral, parasitic, or fungal in either eye at the baseline visit.
4. Contraindication to pupillary dilation in either eye.
5. Uncontrolled systemic disease.
6. Any condition (including inability to read visual acuity charts and language barriers) which precludes subjects ability to comply with the study requirements including the completion of the study.
7. Subject has a condition or is in a situation which the investigator's opinion may put the subject at significant risk, may confound the study results or may interfere significantly with the subjects participation in the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Male or female at least 50 years of age.
  2. Subjects must have age related macular degeneration with a choroidal neovascular membrane either classic or occult in at least one eye.
  3. Preoperative best corrected visual acuity (BCVA) equal to or greater to 19 letters on the ETDRS diabetic retinopathy study chart (20/400 Snellen).
  4. Media clarity, pupillary dilation and subject cooperation sufficient for accurate OCT and angiographic assessment.
  5. Written and informed consent has been obtained.
  6. Written authorization for the use and release of the health and research study information in the United States of America USA.
  7. Ability to understand the informed consent and willingness to follow study instruction and likely to complete all required visits and procedures.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2011-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
BEST CORRECTED VISUAL ACUITY AFTER TREATMENTS | 3, 6 12, 15, 18 AND 24 MONTHS AFTER ENTRY
  BEST CORRECTED VISUAL ACUITY AFTER TREATMENTS WITH THOSE ON SUPPLEMENTS VERSUS BEST CORRECTED VISUAL ACUITY OF THOSE WHO JUST RECEIVED TREATMENTS

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Olk, MD, Principal Investigator — The Retina Center
Locations (1):
- The Retina Center, St Louis, Missouri, United States

REFERENCES:
- [Derived] Brown GC, Brown MM, Gierhart D, Olk RJ. Prevention Surpasses Treatment: 5-year Follow-Up, Cost-Utility, and Cost-Benefit of Zeaxanthin Therapy for Neovascular Age-Related Macular Degeneration. Ophthalmol Ther. 2023 Oct;12(5):2583-2608. doi: 10.1007/s40123-023-00742-9. Epub 2023 Jul 10. PMID 37430077